CLINICAL TRIAL: NCT06267404
Title: Effectiveness of Iliopsoas Positional Release Versus Conventional Exercises in the Management of Sub-acute Back Pain in Pakistani Population
Brief Title: Effectiveness of Iliopsoas Positional Release Versus Conventional Exercises in the Management of Sub-acute Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: Sindh Institute of Physical Medicine and Rehabilitation (Other)
Responsible Party: Principal Investigator, Iram Iqbal Shamsi, Principle investigator, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IShamsi
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Back Pain
Keywords: Back ache; Manual therapy; Soft tissue techniques
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iliopsoas positional release (Experimental): Group A (Iliopsoas positional release group) Positional release therapy will be administered on both Iliopsoas muscles, three sets on each side with 30 seconds hold on tender point. A rest of 15 seconds will be given between all sets.
  Interventions: Other: Iliopsoas Positional release therapy
- Conventional therapy (Active Comparator): Group B (Conventional therapy) Conventional Physical therapy i.e. Ultrasonic therapy 3 min 1 MHz, TENS 10 min, hot pack for 10 min and back strengthening exercises.
  Interventions: Other: Conventional exercises

INTERVENTIONS:
Other: Iliopsoas Positional release therapy — Group A(Iliopsoas Positional release group) Patient supine, with both hips are fully extended .Find a Tender point in Iliopsoas muscle, at the initiation of pain Passively try combination of flexion Adduction/Abduction medial or lateral rotation at hip joint and stop where pain start to diminished. Hold this position of relief for 30 seconds until minimum of 75% of relief is achieved. Apply three times, than passively take lower limb in extension. Administered on both limbs.
  Other Names: Strain Counter-strain therapy
  Arms: Iliopsoas positional release
Other: Conventional exercises — Group B (conventional Physical therapy) For Ultra sonic therapy Patient prone lying, Aqua-sonic gel is applied to lumbosacral area and ultrasonic head is moved in circular motion. For TENS Electrodes are placed in crossed pattern, Paravertebral at L1 and L5 (Box Pattern)with circuit crossing at L3 and current is applied for 10 minutes, Hot pack which is kept in hydro-collateral at 70°C and 75°C is, wrapped in several towel layers, applied for 10 minutes.
  Other Names: conventional physical therapy treatment
  Arms: Conventional therapy

SUMMARY:
Recommended treatment for chronic non-specific LBP is exercise therapy, behavioral therapy including pain management, or a combination of these; There is not enough evidence to establish recommendations for which one is the most appropriate.

The primary objective of this study is to explore the effects of Ilio-psoas Release on Sub-acute back pain, ROM & functional disability

DETAILED DESCRIPTION:
Following the screening, participants will be randomized to receive the experimental or the controlled treatment in a1:1 ratio. Computer-generated random numbers will be used for Randomization. After obtaining the basic information, a unique code will be provided to each included patient. The outcome assessor will be blinded to the type of treatment. Patients and investigator could not be blinded due to the nature of treatment.

Group "A "(experimental group) will receive Positional Release Technique on Painful Iliopsoas(Both if Necessary) Group "B" (control group) will receive conventional physical therapy treatment consisting of hot pack, TENS, Ultra Sound along with back strengthening exercises.

All patients will be Assessed for Pain , ROM and Functional Activities before and after treatment sessions.

Visual Analogue Scale(VAS) and Modified Schober Test will be used for pain and ROM respectively. Roland-Morris Questionnaire (RMQ) will be used for functional activities.

ELIGIBILITY:
Inclusion Criteria:

* Sub-acute (pain for > 1.5 month)
* Age 18-40 years
* Willing to participate
* Both gender will be recruited.

Exclusion Criteria:

* Any history related to spinal surgery
* Previous administration of epidural injections
* LBP due to specific pathology
* Neurological deficits (like stroke)
* Clinical disorder contraindicated to exercise

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
VAS Visual Analogue Scale VAS Visual Analogue Scale | Baseline and After Four weeks of Treatment
  The visual analogue scale is used for measurement of pain intensity. It is a continuous scale. It comprises a horizontal or vertical 10 centimeters or 100 millimeters line. The higher scores shows higher pain intensity and lower scores shows lower pain intensity.
Modified Schober's test | Baseline and After Four weeks of Treatment
  It is used during physical examination to assess the lumbar range of movement. It is highly co-related with lumbar range of movement measured through radiograph. Higher score reflect better range of motion of Spine.

SECONDARY OUTCOMES:
Roland-Morris Disability Questionnaire | Baseline and After Four weeks of Treatment
  The Roland-Morris is a 24-item self-report questionnaire about how low-back pain affects functional activities.0 Score means No disability and score 24 means severe disability.
  Each question is worth one point so scores can range from 0 (no disability) to 24 (severe disability).Reduction in score shows Improvement

CONTACTS AND LOCATIONS:
Overall Officials: Iram I Shamsi, M.Phil., Principal Investigator — Sind Institute of Physical Medicine & Rehabilitation; Basit Ansari, PhD, Study Chair — University of Karachi; Aftab A Mirza Baig, PhD, Study Director — IQRA University; Syed A Ali, PhD, Study Director — Government degree Science & commerce college
Locations (1):
- Sindh Institute of Physical Medicine and Rehabilitation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brennan GP, Fritz JM, Hunter SJ, Thackeray A, Delitto A, Erhard RE. Identifying subgroups of patients with acute/subacute "nonspecific" low back pain: results of a randomized clinical trial. Spine (Phila Pa 1976). 2006 Mar 15;31(6):623-31. doi: 10.1097/01.brs.0000202807.72292.a8. PMID 16540864
- [Result] Pfieffer ML. Evaluating and managing low back pain in primary care. Nurse Pract. 2019 Aug;44(8):40-47. doi: 10.1097/01.NPR.0000574664.42110.77. PMID 31335502
- [Result] Ehrlich GE. Back pain. J Rheumatol Suppl. 2003 Aug;67:26-31. PMID 12926648
- [Result] Bardin LD, King P, Maher CG. Diagnostic triage for low back pain: a practical approach for primary care. Med J Aust. 2017 Apr 3;206(6):268-273. doi: 10.5694/mja16.00828. PMID 28359011
- [Result] Krismer M, van Tulder M; Low Back Pain Group of the Bone and Joint Health Strategies for Europe Project. Strategies for prevention and management of musculoskeletal conditions. Low back pain (non-specific). Best Pract Res Clin Rheumatol. 2007 Feb;21(1):77-91. doi: 10.1016/j.berh.2006.08.004. PMID 17350545